CLINICAL TRIAL: NCT04209998
Title: New Oxymetry Indices in Critical Limb Ischemia (French Original Title is "Nouveaux Indices Oxymétriques Chez Les Patients Vus Pour Suspicion d'Ischémie Critique du membrE inférieur")
Brief Title: New Oxymetry Indices in Critical Limb Ischemia
Acronym: NOVICE
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019-A02619-48
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Critical Limb Ischemia
Keywords: transcutaneous oximetry; oxygen; peripheral artery disease; follow-up
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease | interventions — Blood Gas Monitoring, Transcutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: transcutaneous oximetry — Analysis of transcutaneous oximetry (Tcpo2) in terme of variability at rest and of response to oxygen inhalation
  Other Names: oxygen inhalation

SUMMARY:
Transcutaneous oxygen tension (TcpO2) at rest, sensitized by oxygen inhalation tests, is widely applied for the evaluation of chronic critical limb ischemia (CLI). If foot TcpO2 measurements are good prognostic factors of the risk of amputation or the probability of wound healing without amputation, they have never proven their hability to estimate the risk of death in patients with critical limb ischemia. On the one hand, studies have considered only the response observed on legs without considered the thoracic variations. On the other hand, the variability of the TcpO2 signal has never been analyzed as a prognostic factor.

The objective of the NOVICE study is therefore to assess, first, whether the variability of resting TcPO2 values at thoracic probe as well as at affected limb probe is a morbidity-mortality prognostic factor and secondly, to evaluate during the oxygen tests, if the measurement of the amplitude of the distal responses in ischemic zone compared to the response observed in thoracic probe is a prognostic factor of morbi-mortality.

DETAILED DESCRIPTION:
This is an ambispective (both retrospective and prospective) cohort study in which any major patient, referred for resting (transcutyaneous oxygen pressure = TcpO2) for suspicion of critical limb ischemia, is included retrospectively and prospectively from November 2018 to October 2020. Tcpo2 recording are analysed to determine specific parameters (signal variability and response top oxygen). A morbidity-mortality follow-up is carried out between 12 and 15 months after the Tcpo2 measurement. A Kaplan Mayer study of these indices against MALE (major adverse lower limb events ) and MACE(Major adverse cardiovascular events) will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of Critical limb ischemia
* Reffered for Tcpo2 Absence of rebuttal to the use of the data by the patients

Exclusion Criteria:

* No available tcpo2 recording
* Rejection of the follow up by the patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for Tcpo2 recording for suspicion of critical limb ischemia.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 12 months
  presence of MACE (major adverse cardiovascular event) following the oximetry test

SECONDARY OUTCOMES:
Morbidity | 12 moths
  presence of MALE (major adverse lower limb event) following the oximetry test
Mortality (intermediate analysis) | 6 months minimal follow-up
  Mortality all causes (intermediate analysis prior to Covid interference)

CONTACTS AND LOCATIONS:
Overall Officials: ABRAHAM Pierre, MD PhD, Principal Investigator — University Hospital in Angers
Locations (1):
- Centre hospitalier universitaire, Angers, France